CLINICAL TRIAL: NCT06919211
Title: Outcomes of Perfluorocarbon Liquid vs. Posterior Retinotomy During Pars-plana Vitrectomy for The Surgical Repair of Rhegmatogenous Retinal Detachment
Brief Title: Perfluorocarbon Liquid vs. Posterior Retinotomy During Pars-plana Vitrectomy for Rhegmatogenous Retinal Detachment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer of Ophthalmologyو Department of Ophthalmology, Faculty of Medicine, Benha University, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ophth._20/2024Med.Research
Record Dates: First submitted 2025-03-29; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Rhegmatogenous Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perfluorocarbon Liquid Group (Experimental)
  Interventions: Procedure: Perfluorocarbon Liquid vs. Posterior Retinotomy during Pars-plana Vitrectomy for The Surgical Repair of Rhegmatogenous Retinal Detachment
- Posterior Retinotomy Group (Experimental)
  Interventions: Procedure: Perfluorocarbon Liquid vs. Posterior Retinotomy during Pars-plana Vitrectomy for The Surgical Repair of Rhegmatogenous Retinal Detachment

INTERVENTIONS:
Procedure: Perfluorocarbon Liquid vs. Posterior Retinotomy during Pars-plana Vitrectomy for The Surgical Repair of Rhegmatogenous Retinal Detachment — This study compares outcomes of perfluorocarbon liquid (PFCL) versus posterior retinotomy (PR) during Pars plana vitrectomy (PPV) for Rhegmatogenous retinal detachment (RRD), focusing on anatomical success, visual acuity, intraocular pressure (IOP), and complications

SUMMARY:
Purpose To evaluate the outcomes of perfluorocarbon liquid (PFCL) versus posterior retinotomy (PR) during Pars plana vitrectomy (PPV) for Rhegmatogenous retinal detachment (RRD), focusing on anatomical success, visual acuity, intraocular pressure (IOP), and complications.

Methods This is a prospective randomized controlled trial that included 58 eyes with RRD, divided into Group A (PFCL, n = 29) and Group B (PR, n = 29). Preoperative assessments included best-corrected visual acuity (BCVA), IOP, axial length, lens status, macula status, and PVR grade. Outcomes were evaluated at 1 week, 1 month, 2 months, and 3 months postoperatively. Primary outcomes included retinal reattachment rates and the number of operations; secondary outcomes included BCVA, IOP changes, complications like cataract development, retinal redetachment, epiretinal membrane (ERM) formation, and single-surgery success.

ELIGIBILITY:
Inclusion criteria:

A clear diagnosis of primary RRD requiring surgery, 18 years or older, The potential to return for follow-up visits for at least 6 months post-surgery.

Exclusion criteria:

When presented with tractional or exudative retinal detachment, had surgery on the affected eye in the past, presented with severe eye disorders like advanced glaucoma or endophthalmitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Retinal reattachment rates | One month, Two months, and Three Months
Number of operations | One month, Two months, and Three Monthes

SECONDARY OUTCOMES:
Best-corrected visual acuity (BCVA) | One month, Two months, and Three Monthes
Intraocular pressure (IOP) | One month, Two months, and Three Monthes
Complications like cataract development, retinal redetachment, epiretinal membrane (ERM) formation, and single-surgery success | One month, Two months, and Three Monthes

CONTACTS AND LOCATIONS:
Locations (1):
- Ebsar Eye Center, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vo LV, Ryan EH, Ryan CM, Shah GK, Gupta OP, Capone A Jr, Eliott D, Yonekawa Y, Bhavsar AR, Emerson MV, Jones JM, Emerson GG. Posterior Retinotomy vs Perfluorocarbon Liquid to Aid Drainage of Subretinal Fluid During Primary Rhegmatogenous Retinal Detachment Repair (PRO Study Report No. 10). J Vitreoretin Dis. 2020 Aug 12;4(6):494-498. doi: 10.1177/2474126420941372. eCollection 2020 Nov-Dec. PMID 37007660
- [Background] Vidne O, Blum Meirovitch S, Rabina G, Abd Eelkader A, Prat D, Barequet D, Moisseiev J, Moisseiev E. Perfluorocarbon Liquid Vs. Subretinal Fluid Drainage during Vitrectomy for the Primary Repair of Rhegmatogenous Retinal Detachment: A Comparative Study. Curr Eye Res. 2018 Nov;43(11):1389-1394. doi: 10.1080/02713683.2018.1490436. Epub 2018 Jul 9. PMID 29912572
- [Derived] Mohamed Elsayed Saad E, Elbadry Mohammed Mohammed H, Mohamed-Aly Ibrahim M, Hassan Salama Selim O, Mostafa Elsayed Abdelhafeez S, Mohammed Sakr A, Mohamed Abo Elftouh Elsalhy F, Abdelmohsen Ali Ayoub A, Abdelsamea Alazab E, Tharwat E, Gamal El Sayed Mostafa T. Outcomes of perfluorocarbon liquid vs. posterior retinotomy as adjuncts during pars-plana vitrectomy for the surgical repair of rhegmatogenous retinal detachment: a randomized clinical trial. BMC Ophthalmol. 2025 Aug 19;25(1):476. doi: 10.1186/s12886-025-04271-w. PMID 40830767
- See also: Related Info — https://eyewiki.org/Retinal_Detachment
- Available data/document: Study Protocol — https://eyewiki.org/Retinal_Detachment